CLINICAL TRIAL: NCT00644215
Title: Comparison of Subconjunctival 5-FU Injection and Mitomycin C for Treatment of Early Bleb Failure, a Randomized Clinical Trial
Brief Title: Comparison of Subconjunctival 5-Fluorouracil (FU) Injection and Mitomycin C for Treatment of Early Bleb Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Mohammad pakravan ,M.D, ophthalmic research center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8662
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Bleb
Keywords: injected bleb; mitomycin drop; 5-Fu injection; early bleb failure
MeSH Terms: conditions — Blister | interventions — Fluorouracil; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 5-FU injection has been done
  Interventions: Drug: 5-FU and Mitomycin
- 2 (Experimental): Mitomycin drop has been administrated
  Interventions: Drug: 5-FU and Mitomycin

INTERVENTIONS:
Drug: 5-FU and Mitomycin — * 5-FU injection 5mg
  * Mitomycin drop 0.02%

SUMMARY:
purpose : to evaluate and compare the effectiveness and complication of 5-FU injections and MMC drop in management of early bleb failure .

Design:Randomized clinical trial Methods:Patients with low injected bleb in first month after filtering or combined surgery with MMC which don't respond to high frequent topical steroids and removal of releasable sutures will be randomize to either 5-FU injection or Mitomycin drop 0.02%.For each patient slit photograph in first day of recruiting,first two weeks and first and third month will be obtained.Patients will follow for at least 3 months and IOP ,bleb configuration will check as primary outcome measures.Preoperative and postoperative data,complications,and the need for further surgical procedures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low,injected bleb in first month after trabeculectomy or combined trabeculectomy&phaco which not respond to high frequent topical steroids or removal of releasable sutures

Exclusion Criteria:

* Injected bleb due to complications of surgery such as button hole formation
* Injected bleb due to blebitis
* Bleb leakage
* Flat AC
* Pregnant or nursing mothers
* Injected bleb after bleb reconstruction

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Iop and Bleb height,extent and vascularity | At least in 3 months of follow up

SECONDARY OUTCOMES:
complication of 5-FU injection or Mitomycin drop in treatment of early bleb failure

CONTACTS AND LOCATIONS:
Locations (1):
- labbafinejad Medical Center,Tehran-Boostan 9 St,Pasdaran Ave,, Tehran, Tehran Province, Iran